CLINICAL TRIAL: NCT02980588
Title: Comparing SGC and Conventional Empiric Treatment for Glucose Control in Critically Ill Patients With Sepsis in ICU
Brief Title: The Effects of SGC on Glucose Control in Critically Ill Patients With Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Chun Pan, Dcotor, Southeast University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zhongda-ICU-SGC
Record Dates: First submitted 2016-11-17; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Sepsis; Hyperglycemia; Critical Illness
MeSH Terms: conditions — Sepsis; Hyperglycemia; Critical Illness

ARMS (1):
- conventional empirical glycemic control (Other): the patients' blood glucose is controlled by physician according to their experience through insulin subcutaneous injection or insulin continuous infusion whose dosage is determinated by the physician.
  Interventions: Device: SGC directed glycemic control

INTERVENTIONS:
Device: SGC directed glycemic control — the patients' blood glucose is controlled by SGC system through insulin continuous infusion whose dosage is determinated by SGC

SUMMARY:
Poorly glycemic control in critically ill patients can increase their mortality, while safe and efficient glucose control is laborious and time-consuming. The Space Glucose Control which is installed with eMPC(enhanced Model Predictive Control) can get the blood glucose target range safely and effectively through regulating insulin dose rate, and decrease the glucose variability. This study is a random controlled trial involving the patients with sepsis in intensive care unit in order to evaluate the difference of safety and efficacy of blood glucose control between SGC directed and conventional treatment. At last, the trial results can determine whether the Space Glucose Control can control blood glucose safely and effectively in the patients with sepsis in intensive care units.

DETAILED DESCRIPTION:
Design: The study was conducted as a single-centre, open randomized controlled, parallel trial.

Study population: Adult general ICU patients with sepsis and assumed to require at least 3 days of intensive care were recruited. Patients fulfilling the inclusion criterion of glucose≥9.0 mmol/L were randomly assigned using serially numbered to either the intervention group (BG control by SGC) or the control group (conventional empiric BG management). The both group aim to establish the BG levels 5.8-8.9mmol/L.

Study protocol: BG measurements were performed using glucometer to test the fingertip capillary blood sample for the BG levels. As for patients with shock or required vasopressor, arterial BG was sampled to measure through the glucometer. Insulin was infused intravenously applying the standard perfusor of the ICU. Average glucose, glucose variability, SOFA score, APACHE II score, and HLA-DR were recorded. All trial-related activities were carried out until the end of the patient's ICU stay, or for a period of 72 hours. Meanwhile, enteral and parenteral nutrition was administrated to patients according to their condition.

Statistical analysis was performed on an intention-to-treat basis. The percentage of values in the target range (5.8-8.9mmol/L) was defined as primary end point for the assessment of glucose control. Data are reported as mean±SD values if not otherwise indicated. Data analysis was performed using SPSS19.0.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the ICU
2. At least one BG measurement 9.0mmol/L or higher
3. Expected to stay in ICU ≥3 days;
4. critically ill patients with sepsis
5. SOFA score≤2

Exclusion Criteria:

1. Aged < 18 years;
2. Admitted because of diabetic ketoacidosis or nonketotic hyperosmolar state
3. Pregnant
4. In a state in which death was perceived as imminent
5. Without written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
glucose variability | up to 3days
  mean blood glucose, standard deviation (SD) for the mean glucose,minimum and maximum glucose levels

SECONDARY OUTCOMES:
HLADr | up to 3days